CLINICAL TRIAL: NCT00420004
Title: A Study of the Effects of LY2216684, a Selective Norepinephrine Reuptake Inhibitor (NERI), in the Treatment of Major Depression
Brief Title: A Study for Participants With Major Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11174; H9P-MC-LNBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY2216684 (Experimental): LY2216684: flexible dose of 3, 6, 9, or 12 milligrams (mg), tablets, administered orally, once daily for 8 weeks.
  For the first week of treatment, participants received a starting dose of 3 mg/day. Then, based on tolerability, for the next 7 weeks, the dose could remain at 3 mg/day; it could be increased 3 mg at a time (scheduled visit) to a maximum dose of 12 mg/day; or it could be decreased 3 mg at any time (scheduled or unscheduled visits) to a minimum dose of 3 mg/day.
  All participants were required to take an equal number of tablets (2) and capsules (2) per day. Therefore, participants on 3 mg/day and 6 mg/day of LY2216684 also received 1 LY2216684-matching placebo tablet + 2 escitalopram-matching placebo capsules. Participants on 9 mg/day and 12 mg/day of LY2216684 also received 2 escitalopram-matching placebo capsules.
  Interventions: Drug: LY2216684; Drug: Placebo
- Placebo (Placebo Comparator): Placebo: tablet and capsule equivalents to LY2216684 and escitalopram, respectively, administered orally, once daily for 8 weeks.
  Interventions: Drug: Placebo
- Escitalopram (Active Comparator): Escitalopram: flexible dose of 10 or 20 milligram (mg), capsules, administered orally, once daily for 8 weeks.
  For the first week of treatment, participants received a starting dose of 10 mg/day. Then, based on tolerability, for the next 7 weeks, the dose could remain at 10 mg/day; it could be increased up to a maximum dose of 20 mg/day; or it could be decreased back to 10 mg/day.
  All participants were required to take an equal number of tablets (2) and capsules (2) per day. Therefore, participants on 10 mg/day of escitalopram also received 1 escitalopram-matching placebo capsule + 2 LY2216684-matching placebo tablets. Participants on 20 mg/day of escitalopram also received 2 LY2216684-matching placebo tablets.
  Interventions: Drug: Placebo; Drug: Escitalopram

INTERVENTIONS:
Drug: LY2216684 — 3-mg and 6-mg tablets
  Other Names: Edivoxetine
  Arms: LY2216684
Drug: Placebo
Drug: Escitalopram — 10-mg capsules
  Other Names: Lexapro®; Cipralex®
  Arms: Escitalopram

SUMMARY:
This is a study to assess the safety and effectiveness of LY2216684 compared to placebo in treating adults with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for major depressive disorder (MDD) without psychotic features.
* Have education level and a degree of understanding such that the participant can communicate with the site study personnel.
* Judged to be reliable and agree to keep all appointments for clinic visits, tests, and procedures, including venipuncture, and examinations required by the protocol.

Exclusion Criteria:

* Have had any additional, ongoing psychiatric condition other than major depression or dysthymia that was considered the primary diagnosis within 6 months of the first study visit.
* Have a lifetime history of Bipolar I or II Disorder, psychotic disorder, or a factitious disorder.
* Are judged to be at high risk for imminently harming themselves or others.
* Have a serious medical illness, including any cardiovascular, hepatic, respiratory, hematologic, endocrinologic, neurologic disease, or clinically significant laboratory or electrocardiogram (ECG) abnormality. Clinically significant lab abnormalities are those which, in the judgment of the investigator, indicate a serious medical problem or require intervention.
* Have any diagnosed medical condition which could be exacerbated by treatment with LY2216684, including hypertension, increased heart rate, arrhythmias, heart disease, narrow angle glaucoma, or urinary hesitancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2006-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Allentown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Media, Pennsylvania
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lasi

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 701 participants were included in a screening/washout period (from 3 to 30 days in duration) prior to group assignments; 232 participants discontinued during this period, and 469 participants were randomized. There was an 8-week Double-blind Phase followed by a 1-week Discontinuation Phase after abrupt discontinuation of treatment.
Groups:
- LY2216684: LY2216684: flexible dose of 3, 6, 9, or 12 milligrams (mg), tablets, administered orally, once daily for 8 weeks
- Escitalopram: Escitalopram: flexible dose of 10 or 20 mg, capsules, administered orally, once daily for 8 weeks
Period: Overall Study
Arm/Group | LY2216684 | Placebo | Escitalopram
Started | 269 | 138 | 62
Received at Least 1 Dose of Study Drug | 249 (Participants who received >=1 dose of study drug and had baseline and post-baseline data available) | 122 (Participants who received >=1 dose of study drug and had baseline and post-baseline data available) | 54 (Participants who received >=1 dose of study drug and had baseline and post-baseline data available)
Completed | 140 | 67 | 30
Not Completed | 129 | 71 | 32
Not completed — Adverse Event | 4 | 1 | 1
Not completed — Lack of Efficacy | 5 | 4 | 1
Not completed — Lost to Follow-up | 31 | 12 | 10
Not completed — Entry Criteria Not Met | 0 | 1 | 0
Not completed — Physician Decision | 14 | 4 | 2
Not completed — Protocol Violation | 5 | 4 | 3
Not completed — Withdrawal by Subject | 67 | 42 | 14
Not completed — Sponsor Decision | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2216684 | Placebo | Escitalopram | Total
Number analyzed (Participants) | 269 | 138 | 62 | 469
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.64 (10.21) | 37.54 (10.97) | 34.32 (9.66) | 36.60 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 65 | 22 | 217
  Male | 139 | 73 | 40 | 252
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 30 | 21 | 8 | 59
  African | 6 | 5 | 0 | 11
  Hispanic | 23 | 7 | 4 | 34
  Native American | 1 | 0 | 0 | 1
  West Asian (Indian subcontinent) | 209 | 105 | 50 | 364
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 23 | 8 | 70
  Romania | 7 | 4 | 1 | 12
  India | 208 | 105 | 50 | 363
  Mexico | 15 | 6 | 3 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in the 17-item Hamilton Depression Rating Scale (HAMD-17) Total Score
Description: The HAMD-17 is a 17-item assessment used to assess the severity of depression and its improvement during the course of therapy. Each item was evaluated and scored using either a 5-point scale of 0 (not present/absent) to 4 (very severe) or a 3-point scale of 0 (not present/absent) to 2 (marked). Higher scores indicate greater symptom severity. The total score was the sum of the scores from HAMD-17 Items 1 through 17 and ranged from 0 (not at all depressed) to 52 (severely depressed). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Baseline, Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline HAMD-17 value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 248 | 122 | 54
units on a scale | -13.2 (0.53) | -12.6 (0.74) | -14.7 (1.14)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.494, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline to Week 8 in Maier-Philipp Subscale of the 17-item Hamilton Depression Rating Scale (HAMD-17)
Description: The HAMD-17 is a 17-item assessment used to assess the severity of depression and its improvement during the course of therapy. Each item was evaluated and scored using either a 5-point scale of 0 (not present/absent) to 4 (very severe) or a 3-point scale of 0 (not present/absent) to 2 (marked). Higher scores indicate greater symptom severity. The Maier-Phillip subscale of the HAMD-17 represents the 6 "core" symptoms of depression (items: 1=depressed mood, 2=feelings of guilt, 7=work and activities, 8=retardation, 9=agitation, 10=anxiety/psychic). The subscale scores range from 0 (normal) to 24 (severe). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Baseline, Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline Maier-Philipp subscale value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 248 | 122 | 54
units on a scale | -6.7 (0.26) | -6.2 (0.36) | -7.6 (0.55)

3. Secondary Outcome: Response and Remission Rates
Description: A participant meets response criteria if there is at least a 50% reduction in the 17-item Hamilton Depression Rating Scale (HAMD-17) total score from baseline to the last observation carried forward (LOCF) endpoint visit. A participant meets remission criteria if the HAMD-17 total score is less than or equal to 7 at the LOCF endpoint visit. The percent of participants meeting criteria is summarized. HAMD-17 is a 17-item assessment used to assess the severity of depression and its improvement during the course of therapy. Each item was evaluated and scored using either a 5-point scale of 0 (not present/absent) to 4 (very severe) or a 3-point scale of 0 (not present/absent) to 2 (marked). Higher scores indicate greater symptom severity. The total score was the sum of the scores from HAMD-17 Items 1 through 17 and ranged from 0 (not at all depressed) to 52 (severely depressed).
Time Frame: Baseline, up to Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline HAMD-17 total score value. Last observation carried forward (LOCF) methodology was used.
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 248 | 122 | 54
percentage of participants
  Response | 54.0 | 48.4 | 53.7
  Remission | 38.7 | 31.1 | 42.6

4. Secondary Outcome: Clinical Global Impression of Improvement Score at Week 8
Description: The Clinical Global Impression of Improvement (CGI-I) scale measures the clinician's perception of participant improvement at the time of assessment compared with the start of treatment. Scores range from 1 (very much improved) to 7 (very much worse). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, and treatment-by-visit.
Time Frame: Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline CGI-I value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 247 | 122 | 53
units on a scale | 2.2 (0.09) | 2.3 (0.12) | 2.0 (0.19)

5. Secondary Outcome: Change From Baseline in Hamilton Anxiety Rating Scale (HAMA) Total Score up to Week 8 Endpoint
Description: The HAMA is a 14-item assessment used to assess the severity of anxiety. The investigator talked to the participant about the symptoms he or she experienced during the previous week. Each item was scored using a 5-point scale (0=not present to 4=very severe). The total score of HAMA ranged from 0 (normal) to 56 (severe). Least Squares (LS) means were adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, up to Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline HAMA value. Last observation carried forward (LOCF) methodology was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 212 | 106 | 44
units on a scale | -9.7 (0.62) | -9.6 (0.82) | -11.6 (1.19)

6. Secondary Outcome: Change From Baseline on the 36-item Short-Form (SF-36) Health Status Survey Mental and Physical Components up to Week 8 Endpoint
Description: The SF-36 Health Status Survey is a generic, health-related scale assessing a participant's quality of life on 8 domains: general health (GH), physical functioning (PF), role-physical, role-emotional, social functioning, bodily pain, vitality, and mental health. Each domain is scored by summing the individual items (GH [range: 5-25]; PF [range: 10-30]; role-physical [range: 4-8]; role-emotional [range: 3-6]; social functioning [range: 2-10]; bodily pain [range: 2-11]; vitality [range: 4-24]; mental health [range: 5-30]) and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning. Two summary scores (mental component and physical component scores) were constructed based on the 8 SF-36 domains. Mental component summary and physical component summary scores range from 0 to 100 (higher scores indicate better health status).
Time Frame: Baseline, up to Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline SF-36 Health Status Survey value. Last observation carried forward (LOCF) methodology was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 192 | 99 | 41
units on a scale
  Mental Component Summary | 13.4 (13.1) | 12.6 (13.9) | 12.4 (12.4)
  Physical Component Summary | 4.17 (9.00) | 2.37 (8.26) | 2.74 (7.65)

7. Secondary Outcome: Change From Baseline in Quick Inventory of Depressive Symptomatology Total Score up to Week 8 Endpoint
Description: The Quick Inventory of Depressive Symptomatology is a 16-item participant-rated measure of depressive symptomatology. There were 4 possible answers per question that are specific to the question; each question (Q) was scored 0 (no problems) to 3 (increased symptoms). The total score was the sum of the highest number from Q1-4, number from Q5, highest number from Q6-9, total for Q10-14, and the highest number from Q15-16. The total score ranges from 0 to 27 with higher scores indicative of greater severity of depression. Least Squares (LS) means were adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, up to Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline Quick Inventory of Depressive Symptomatology value. Last observation carried forward (LOCF) methodology was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 198 | 103 | 42
units on a scale | -10.2 (0.54) | -8.3 (0.71) | -11.6 (1.04)

8. Secondary Outcome: Change From Baseline in Beck Scale for Suicide Ideation up to Week 8 Endpoint
Description: Beck Scale for Suicide Ideation (BSI) is a 21-item participant-completed questionnaire designed to assess severity of suicidal ideation in adults and adolescents. The BSI total score is calculated as the sum of the responses (rated from 0 to 2 in terms of severity) to the first 19 items of the BSI scale. The BSI total score ranges from 0 to 38, with a higher score indicating a higher degree of suicide ideation.
Time Frame: Baseline, up to Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline BSI value. Last observation carried forward (LOCF) methodology was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 245 | 122 | 51
units on a scale | -0.90 (3.39) | -0.54 (2.14) | -0.78 (2.16)

9. Secondary Outcome: Change From Baseline in Modified Overt Aggression (OAS-M) Scale up to Week 8 Endpoint
Description: OAS-M is a clinician-administered semistructured interview designed to assess various manifestations of aggressive behavior. Final scores are rated on 3 scales: Aggression (Agg), Irritability (Irrt), Suicidality (Suic). Agg scale has 4 subscales: Verbal Assault (Aslt), Aslt Against Objects, Aslt Against Others, Aslt Against Self; each item is scored 0-5, multiplied by the frequency of the behavior, then summed together. Agg total score is the weighted sum of the subscale scores (weights: 1=Verbal Aslt, 2=Aslt Against Objects, 3=Aslt Against Others, 4=Aslt Against Self). The Irrt scale has 2 subscales: Global Irrt, Subjective Irrt. Suic scale has 3 subscales: Suicidal Tendencies, Intent of Attempt, Lethality of Attempt. The 2 Irrt and 3 Suic subscales are rated on 6 or 7 point scales from 0=none/not at all to 6/7=very extreme. The total score ranges from 0-10 for the Irrt scale and 0-16 on the Suic scale. Least Squares means were adjusted for treatment, investigator, and baseline s
Time Frame: Baseline, up to Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline OAS-M value. Last observation carried forward (LOCF) methodology was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 227 | 113 | 47
units on a scale
  Aggression total score | -4.1 (0.52) | -4.2 (0.71) | -3.9 (1.06)
  Irritability total score | -1.0 (0.10) | -0.9 (0.14) | -1.0 (0.20)
  Suicidality total score | -0.2 (0.04) | -0.2 (0.05) | -0.2 (0.08)

10. Secondary Outcome: Change From Baseline in Arizona Sexual Experiences Scale up to Week 8 Endpoint
Description: The Arizona Sexual Experiences Scale (ASEX) is used to assess sexual functioning in both males and females. The ASEX total score for the male and female version is calculated as the sum of the responses (rated from 1 [extremely] to 6 [no/never]) to the 5 items of the ASEX scale. Total scores ranged from 5 to 30 with higher scores indicating greater sexual dysfunction.
Time Frame: Baseline, up to Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline ASEX value. Last observation carried forward (LOCF) methodology was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 219 | 109 | 43
units on a scale | -2.68 (6.65) | -1.69 (6.35) | -1.65 (7.43)

11. Secondary Outcome: Change From Baseline in Insomnia Severity Index up to Week 8 Endpoint
Description: The Insomnia Severity Index (ISI) is a brief self-report instrument measuring the participant's perception of his or her insomnia. The ISI score is calculated as the sum of the responses to the 7 items of the ISI scale. Each item is rated on a 0 to 4 scale and the total score ranges from 0 to 28 with a higher score suggesting more severe insomnia.
Time Frame: Baseline, up to Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline ISI value. Last observation carried forward (LOCF) methodology was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 227 | 113 | 45
units on a scale | -7.53 (7.57) | -7.44 (7.73) | -8.02 (7.72)

12. Secondary Outcome: Change From Baseline to Week 8 in Fatigue Severity Scale
Description: Fatigue Severity Scale (FSS) is a 9-item measure of fatigue severity. Each item is scored by the participant on a scale of 1 ("Disagree") to 7 ("Agree"), with a higher score indicating a stronger agreement with the item statement regarding the participant's fatigue symptoms. The FSS total score ranges from 1 to 7, and is obtained by averaging the responses to the 9 items. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Baseline, Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline FSS value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 225 | 109 | 47
units on a scale | -2.0 (0.14) | -1.8 (0.19) | -2.2 (0.29)

13. Secondary Outcome: Pharmacokinetics: Predicted Maximal Concentration of LY2216684 at Steady State (Cmax,ss) at Week 8 Endpoint
Description: Predicted maximal LY2216684 plasma concentrations at steady state (Cmax,ss) are reported, using the dose at the last visit in the study for participants included in the primary efficacy analysis.
Time Frame: Up to 8 weeks
Population: All participants randomized to LY2216684 included in the primary efficacy analysis with a pharmacokinetic (PK) sample at the participants' final study visit.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | LY2216684
Number analyzed (Participants) | 193
nanograms per milliliter (ng/mL)
  3 mg dose: number analyzed (Participants) | 31
  3 mg dose | 10.5 (2.0)
  6 mg dose: number analyzed (Participants) | 52
  6 mg dose | 22.6 (5.4)
  9 mg dose: number analyzed (Participants) | 44
  9 mg dose | 32 (6.4)
  12 mg dose: number analyzed (Participants) | 66
  12 mg dose | 40.6 (9.9)

14. Secondary Outcome: Number of Participants With at Least 1 Serious Adverse Event (Safety and Tolerability)
Description: The number of participants with at least one serious adverse event, regardless of causality is reported cumulatively through Week 8. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Event module.
Time Frame: Baseline through Week 8
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 269 | 138 | 62
Participants | 2 | 1 | 2

15. Secondary Outcome: Change From Baseline to Week 8 in the 21-item Hamilton Depression Rating Scale (HAM-21) Total Score
Description: The HAMD-21 is a 21-item assessment used to measure depression severity. Items were rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score ranging from 0 (not at all depressed) to 60 (severely depressed). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Baseline, Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline HAMD-21 value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 239 | 120 | 52
units on a scale | -13.6 (0.57) | -13.0 (0.79) | -15.0 (1.24)

16. Secondary Outcome: Cognitive Assessment Battery: Change From Baseline in Word List Learning and Delayed Recall Test (WLDRT) up to Week 8 Endpoint
Description: The WLDRT is a test of visual learning and recall. Participants are shown a series of words (commonly used nouns) and asked to say each of the words aloud, then are asked to recall the words and the total number of correct words recalled is recorded (possible score ranged from 0 to 15 words). The process is repeated 3 times. The Word List Learning Test score is calculated as the average number of words recalled during the first 3 trials. After a 30-minute delay, participants are again asked to recall the words, and the total number of correct words remembered after the delay is recorded as the Delayed Recall Test score. The baseline value was the last non-missing value before the first randomized double-blind study drug administration. Least Squares (LS) means were adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, up to week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who have a baseline and at least one post-baseline WLDRT value. Last observation carried forward (LOCF) methodology was used.
Measure: Least Squares Mean (Standard Error); unit: number of correct words
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 207 | 107 | 43
number of correct words
  Word List Learning Test | 0.5 (0.15) | 0.3 (0.19) | 0.3 (0.28)
  Delayed Recall Test: number analyzed (Participants) | 206 | 107 | 43
  Delayed Recall Test | 0.4 (0.19) | 0.2 (0.25) | 0.0 (0.37)

17. Secondary Outcome: Cognitive Assessment Battery: Change From Baseline in Symbol Digit Substitution Test (SDST) up to Week 8 Endpoint
Description: The SDST is an attention-demanding psychomotor component based on the Digit Symbol Substitution Test from the Wechsler Adult Intelligence Scale. The participant is given a symbol/digit code in which each of the digits 1 through 9 is paired with a different symbol. Below the code, a series of symbols selected from those in the code are presented in an irregular order. The participant is instructed to write the number that is appropriate for each symbol in the space below each symbol and to complete as many correct digits as possible within a 90-second test period. For this test, the number of attempts and number of correct digits is collected. The percentage of correct digits is presented based on the number of correct digits divided by the number of attempts, multiplied by 100 (score ranged from 0 to 100% correct). Least squares (LS) means were adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, up to Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline SDST value. Last observation carried forward (LOCF) methodology was used.
Measure: Least Squares Mean (Standard Error); unit: percentage of correct digits
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 182 | 94 | 39
percentage of correct digits | 3.2 (1.12) | 2.5 (1.42) | 2.2 (2.10)

18. Secondary Outcome: Cognitive Assessment Battery: Change From Baseline in Two Digit Cancellation Test up to Week 8 Endpoint
Description: The Two Digit Cancellation Test (2DCT) is a clinical adaptation of the visual search tasks that have been used to investigate cognitive processes involved in attention and visual information processing. For this test, the participant is presented with a piece of paper containing rows of digits. At the top of the page are two target digits. The participant is instructed to examine each row of digits working from top to bottom and left to right crossing off each number that matches either of the two numbers at the top of the page. The number of targets hit, number of errors, and number of times the participant had to be reminded of the task are recorded for the 45-second test. The 2DCT composite cognitive score is calculated as the number of targets hit - number of errors - number of reminders. 2DCT score ranges 0-40 with higher score indicating better cognition. Least squares (LS) means were adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, up to Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline 2DCT value. Last observation carried forward (LOCF) methodology was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 194 | 99 | 49
units on a scale | 0.8 (0.62) | 1.2 (0.83) | 1.0 (1.26)

19. Secondary Outcome: Cognitive Assessment Battery: Change From Baseline in Trail Making A up to Week 8 Endpoint
Description: Trail Making A is a neurocognitive test associated with general brain function. While being timed, the participant is instructed to connect 25 randomly placed circled numbers on a page in numerical sequence without lifting their pencil. If a participant makes a mistake, the mistake is pointed out and the participant must start again from the last correct circle. The total time to complete the task (up to 300 seconds, with a lower value indicating better brain function) is recorded. Least squares (LS) means were adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, up to Week 8
Population: All randomized participants who received at least one dose of double-blind study drug and who had a baseline and at least one post-baseline Trail Making A value. Last observation carried forward (LOCF) methodology was used.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | LY2216684 | Placebo | Escitalopram
Number analyzed (Participants) | 203 | 104 | 43
seconds | -9.9 (2.97) | -11.1 (3.85) | -5.6 (5.68)

ADVERSE EVENTS:
Groups:
- LY2216684 Double Blind Phase: LY2216684: 3, 6, 9, or 12 milligrams (mg) tablets, administered orally with flexible dosing, once daily for 8 weeks
- Placebo Double Blind Phase: Placebo: tablet and capsule equivalents to LY2216684 and escitalopram, respectively, administered orally once daily for 8 weeks
- Escitalopram Double Blind Phase: Escitalopram: 10 or 20 mg capsules, administered orally with flexible dosing, once daily for 8 weeks
- LY2216684 Discontinuation Phase: Included all randomized participants who discontinued LY2216684 treatment
- Placebo Discontinuation Phase: Included all randomized participants who discontinued placebo
- Escitalopram Discontinuation Phase: Included all randomized participants who discontinued escitalopram treatment
Arm/Group | LY2216684 Double Blind Phase | Placebo Double Blind Phase | Escitalopram Double Blind Phase | LY2216684 Discontinuation Phase | Placebo Discontinuation Phase | Escitalopram Discontinuation Phase
Serious Adverse Events (participants affected / at risk) | 2/269 | 1/138 | 2/62 | 0/269 | 1/138 | 0/62
Other Adverse Events (participants affected / at risk) | 70/269 | 26/138 | 19/62 | 3/269 | 2/138 | 2/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2216684 Double Blind Phase (N=269) | Placebo Double Blind Phase (N=138) | Escitalopram Double Blind Phase (N=62) | LY2216684 Discontinuation Phase (N=269) | Placebo Discontinuation Phase (N=138) | Escitalopram Discontinuation Phase (N=62)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2216684 Double Blind Phase (N=269) | Placebo Double Blind Phase (N=138) | Escitalopram Double Blind Phase (N=62) | LY2216684 Discontinuation Phase (N=269) | Placebo Discontinuation Phase (N=138) | Escitalopram Discontinuation Phase (N=62)
Constipation (Gastrointestinal disorders) | 18 (19) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 17 (17) | 6 (6) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 24 (27) | 5 (5) | 7 (7) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 26 (34) | 9 (9) | 7 (7) | 2 (2) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 14 (15) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days